CLINICAL TRIAL: NCT04937010
Title: Efficacy and Safety of Occipital Nerve Stimulation in Trigeminal Autonomic Cephalalgias: A Double-blind, Phase II, Randomized, Controlled Trial
Brief Title: Occipital Nerve Stimulation in Trigeminal Autonomic Cephalgias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Responsible Party: Principal Investigator, Fady Girgis, Physician, Alberta Health Services, Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB21-0839
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Trigeminal Autonomic Cephalgia
Keywords: Occipital Nerve Stimulation
MeSH Terms: conditions — Trigeminal Autonomic Cephalalgias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Industry standard stimulation (Active Comparator): Standard sub threshold stimulation parameters
  Interventions: Procedure: Occipital nerve stimulator implant
- Experimental stimulation (Sham Comparator): Sham stimulation
  Interventions: Procedure: Occipital nerve stimulator implant

INTERVENTIONS:
Procedure: Occipital nerve stimulator implant — Implantation of occipital nerve stimulator and different stimulation parameters

SUMMARY:
The objective of this study is to determine the efficacy of occipital nerve stimulation (ONS) in the treatment of chronic trigeminal autonomic cephalalgias (TACs).

DETAILED DESCRIPTION:
Several open studies and case series have shown improvement in pain scores using ONS specifically for cluster headache, which is the most common of the TACs. However, neuromodulation in the treatment of pain disorders is subject to strong placebo effect and bias, and the lack of controlled studies in this population makes its true efficacy unknown. Therefore, we plan to study ONS in a population of patients with chronic TACs using a double-blind, randomized, controlled, cross-over study. Using sub-threshold stimulation parameters, meaning patients will not know when therapeutic stimulation is active, subjects will rate their pain and quality of life during both therapeutic and sham stimulation periods. Following the cross-over period, all subjects will undergo therapeutic stimulation for 1-year in order to gauge long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Meets ICHD-3 diagnostic criteria for the chronic form of one of the trigeminal autonomic cephalgias (outlined below), as determined by the treating neurologist.
* Failed standard medical management, meaning at least 3 conventional preventative therapies.

Exclusion Criteria:

* Presence of uncontrolled or untreated psychiatric disease
* Presence of medical contraindications to surgery
* Patient does not consent to surgery
* Non-English speaking

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in headache frequency | 6 months
  Change in frequency of headaches

SECONDARY OUTCOMES:
Safety of Occipital Nerve Stimulation | 6 months
  Any adverse events with stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No